CLINICAL TRIAL: NCT04760054
Title: Effects of a Complex, Partnered Martial Arts-based Intervention on Cognitive Function in Comparison to Aerobic Exercise and Attention-control Among Low-active Adults
Brief Title: Effects of a Complex, Partnered Martial Arts-based Intervention on Cognitive Function
Acronym: HUBOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor Sean Mullen, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21174
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Change; Processing, Visual Spatial; Inhibition (Psychology); Working Memory
Keywords: Cognitive Performance; Complex movement
MeSH Terms: conditions — Spatial Processing; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Three groups: One intervention, One Exercise Comparison, One Attentional Control
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be masked to group allocation. Participants will not be masked from knowledge of other group's activities, but will only receive the training from one specific training group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HUBOD martial arts practice (Experimental): Participants will be trained in the Hubod exercise over 5 separate training sessions. Sessions will last approximately 30 minutes, involving a warm up, review of material from the previous session and the learning of the next movement in the HUBOD sequence. Heartrate will be monitored periodically to make sure the intensity of exercise is consistent with mild to moderate cardiovascular exercise as in the active comparator.
  Interventions: Behavioral: HUBOD
- Active Comparator - Stationary Bicycle (Active Comparator): Participants will be given 5 separate sessions, each approximating 30 minutes in duration, of mild to moderate intensity cardiovascular training on a stationary bicycle. Heartrate will be monitored periodically to make sure the intensity of exercise is consistent with mild to moderate exercise as in the Experimental group.
  Interventions: Behavioral: Active Comparator
- Attentional Control Group (Placebo Comparator): Participants will be given 5 separate sessions, each approximating 30 minutes in duration, of watching videos on martial arts training methods and techniques. These sessions will be completely sedentary.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: HUBOD — Participants in the intervention group will attend 5 separate training sessions instructing them in Hubod. The Hubod exercise is a partnered coordination drill involving moves derived from numerous martial arts, most often seen in the Filipino martial art of Kali. Participants will aim to reach a level of comfort and competency in the basic, non-competitive aspects of the Hubod exercise by the end of their participation in this intervention.
  Other Names: Martial Arts Experimental Exercise Group; Hubod Training Group
  Arms: HUBOD martial arts practice
Behavioral: Active Comparator — Participants in the active comparator group will attend 5 separate training sessions. Each session will involve a 5 minute warmup of joint mobilization exercises and mild pedaling on the bicycle before the main effort of continuously using the bicycle for approximately 20 minutes. The session finishes with a 5 minute cooldown period and light stretch. Heartrate will be monitored regularly in order to prevent this exercise exceeding the relative intensity of the Martial Arts intervention group. Participants will be allowed to talk and interact with research assistants in order to keep socialization effects consistent across groups.
  Other Names: Exercise Comparison Group; Stationary Bike Group
  Arms: Active Comparator - Stationary Bicycle
Behavioral: Control Condition — Participants in this group will attend 5 separate training sessions. Each session will involve watching educational videos on martial arts techniques and training methods from a sedentary position. Participants will be allowed to talk and interact with research assistants in order to keep socialization effects consistent across groups.
  Arms: Attentional Control Group

SUMMARY:
The investigators' study is designed to test whether brief exposure to a martial arts-based intervention (a coordinative, partnered training exercise known as "Hubod"), can improve cognitive function to a greater degree than aerobic exercise of a similar intensity.

DETAILED DESCRIPTION:
This three-arm randomized controlled trial will compare the feasibility, and possibly the effects, of a martial arts intervention vs. aerobic exercise vs. an attentional (non-exercise) control condition. The martial arts intervention will consist of a partnered, coordinated sensitivity exercise drawn from south-east Asian martial arts, known as Hubod (also spelt hubud and hubad). Participants will be trained in the fundamental movements of Hubod. Participants will also have the history, cultural significance, risks and purpose of Hubod explained to them throughout the study.

The aerobic exercise comparator group will use a stationary bicycle to match the duration and exercise intensity of the martial arts intervention group, under the supervision of trained research assistants. Participants will also receive information on aerobic exercise and the Physical Activity Guidelines for Americans 2020.

Participants in the Videos Control group will watch educational videos on martial arts, physical fitness and exercise for the same duration as the intervention and exercise comparison groups. All participants, regardless of group, will be assessed for martial arts and exercise experience once at baseline.

All participants will be tested for cognitive performance change. Baseline and follow-up computerized cognitive testing will take place at a specified testing facility and psychosocial questionnaires will be delivered remotely via a Qualtrics-powered survey. After baseline testing, participants will attend 5 sessions, approximately 30 minutes each. Follow-up testing will be administered more than 48 hours post-intervention to minimize established acute adaptive responses to exercise.

The investigators hypothesize the martial arts training intervention group will exhibit a greater increase in performance of cognitive tasks when compared less complex movement patterns involved in the aerobic exercise group or videos control group.

ELIGIBILITY:
Inclusion Criteria:

- Men and Women between the ages of 18-45 years who are low active

Exclusion Criteria:

* Anyone who is physically active (≥30 minutes, 3 or more times/week, for the last 3 months) and/or a regular practitioner of martial arts and/or highly complex coordination drills such as dance performance or contact improvisation (≥30 minutes, 3 or more times/week, for the last 3 months).
* Anyone with serious chronic medical conditions that would preclude them from participating without a physician present, or anyone with a risk of seizure, or anyone having psychiatric and/or neurological disorders.
* Pregnant women.
* Anyone incapable of performing the following movements at a moderate intensity- sitting, standing, kicking, pulling, pushing, bending one's elbows or bending one's knees.
* Anyone who scores 1 or more on the Physical Activity Readiness Questionnaire
* Anyone refusing or unwilling to be randomized into either of the conditions.
* Anyone who cannot commit to both 45 minute testing sessions or the five 30-minute training sessions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Digit Symbol Substitution task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  Processing speed and working memory cognitive task using numbers and symbols. Participants will be presented with multiple rows of symbols, each one corresponding to a number on a 1-9 scale and they will have two minutes to correctly match (in sequential order) as many symbols to their numbers as possible. Performance is computed by adding the number of symbols correctly-matched within the allotted time.
n-2back memory task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  Working memory cognitive task involving a sequence of shapes briefly appearing on a computer screen. If the shape on screen is identical to the shape two stages before, the participant will press the 'match' key. If they are not identical, the participant should do nothing. Performance is derived by the number of correctly-matched shapes in the sequence and calculating the average reaction time across the trials.

SECONDARY OUTCOMES:
Matrix Reasoning Task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  Participants will be required to identify patterns among objects in an incomplete, 3x3 matrix, according to row and column, and to select the correct object that completes the remaining empty box from a list of potential objects. Performance will be assessed from the number of correct responses within the allotted time.
Trail-Making Test | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  The trail-making test is a global cognition and spatial awareness assessment involving two parts. Respondents must complete each part as quickly as possible using a single, continuous pencil-drawn line. For Trails part A, the numbers 1-26 are randomly arranged on a sheet of paper and respondents are required to connect the numbers, in order, using a single pencil line. The pencil is not allowed to leave the paper until the task is complete. The same is true for Trails part B, but the sequence is now numero-alphabetic (1, A, 2, B, 3, C and so on). The task is complete when the participant reaches the end of the sequence. Performance will be measured by how long it takes the participant to complete parts A and B.
Flanker Task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  The Flanker task paradigm assesses inhibition control. The task utilizes pictures and symbols and is delivered using an iPad. Participants will be required to correctly identify, as fast as possible, the direction a central arrow among a set of surrounding arrows that are pointing in either congruent or incongruent directions. Performance will be assessed using average reaction time responses and accuracy across the congruent and incongruent trials. Inhibition percent interference will be calculated using the formula ((incongruent reaction time - congruent reaction time)/congruent reaction time) * 100.

OTHER OUTCOMES:
Perceived Mental Fatigue Questionnaire | Participants will be assessed at baseline and in the week immediately following the two-week intervention period; also delivered immediately prior to and following each of the five intervention training sessions.
  A novel, 7-item assessment of current state of mental fatigue will be used (example items include "My thoughts easily wander," "My thinking requires effort.") The scales response ranges from 1 (not true at all) to 5 (very true) and all items are summed and averaged whereby higher scores indicated greater mental fatigue.
Grip strength task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  A dynamometer will be used to assess grip strength. Under supervision, participants will engage in two trials per hand (unless each trial results in an increasing or identical score, at which point a third trial will be used). The highest score, as well as an average of the two highest scores, will be recorded as measures of grip strength from this task.
Stair-climb task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  To assess mobility, participants will be asked to walk up and down a single 15-step staircase. After explanation and demonstration of the task, participants will be asked to safely descend as quickly as possible, without skipping stairs, running or using the railing for assistance. The same will be asked for participants during stair ascension. Performance will be recorded as total time (seconds) to complete stair ascent and descent.
One-leg balance task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  Balance will be assessed by asking participants to stand on one leg for a maximum of 30 seconds. Participants may not use any assistance and performance will be recorded as balance time (in seconds) without touching the floor or their base leg with their elevated leg.
Dot task | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  Agility will be assessed with a timed, choreographed sequence of steps on a dotted floor mat (positioned in an X-pattern). Performance will be based on how quickly (measured in seconds) they can perform the prescribed, choreographed sequence.
Godin Leisure-Time Exercise Questionnaire | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  This is a 4-item self report assessment of physical activity. Respondents are asked the frequency they engage in strenuous, moderate and mild activity for 15 minutes or more as part of their free time.
Brief Self Control Scale | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  13-item self-reported measure of individual differences in control. Items are scored on a 1-5 likert scale (1 = not at all like me, 5 = Very much like me). Scores are totaled and the mean average calculated to be used in final analysis.
Multidimensional Outcomes Expectations for Exercise Scale | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  The Multidimensional Outcome Expectancies for Exercise Scale (MOEES; Wójcicki, White, & McAuley, 2009) is a 15-item questionnaire that has three subscales: physical outcome expectancies, social outcome expectancies, and self-evaluative outcome expectancies. The MOEES assesses an individual's beliefs or expectations about the benefits of regular exercise. Each question is based on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Each subscale is scored by summing the total items, with higher scores being indicative of higher outcome expectations for exercise.
Exercise Motivations Inventory-2 | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  The Exercise Motivations Inventory-2 will be used to assess the type of reasons one has for participating in an exercise program (and their relative strength). Only subscales with items involving appearance, strength/endurance, nimbleness and positive health will be used. Composite scores will be computed for each subscale by summing and averaging responses.
State Trait Anxiety Inventory | Participants will complete this questionnaire immediately prior and immediately following each of the five intervention training sessions.
  Trait anxiety, or one's disposition to respond with anxiety to situations perceived as threatening will be assessed with the State Train Anxiety Inventory. It comprises 20 items (11 direct worded and 9 reverse worded), and respondents answer according to how they generally feel; responses are provided on a frequency scale ranging from 1 (almost never) to 4 (almost always). Composite scores are computed by summing and averaging items.
Hospitalized Anxiety and Depression Scale | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  The established Hospitalized Anxiety and Depression scale consists of 14 questions, and utilizes a 0 to 3-point Likert scale. Oddly numbered questions comprise the Anxiety subscale and evenly numbered questions comprise the Depression subscale. Six items are reversely coded. The sum of item scores in these questions are the final outcome scores per subscale, with 0-7 considered normal, 8-10 considered borderline abnormal and 11-21 considered abnormal.
Physical Activity Self Regulation Questionnaire | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  A 12-item questionnaire will be used to assess one's usage of self-regulatory strategies that promote physical activity including cognitive and behavioral strategies. Items are scored 1 (Never) to 5 (Very often). Our prior work has determined that this scale is not uni-dimensional across samples. We will therefore use an empirically-driven factor analysis to determine the best set of items to include in the mean composite.
Self-efficacy for overcoming barriers to exercise | Participants will be assessed at baseline and in the week immediately following the two-week intervention period.
  A 13-item questionnaire will be used to assess self-efficacy specific to possible barriers affecting exercise adherence. All items will be answered on a 0-100% Likert scale in increments of 10%. Prior research suggests that this may not be a uni-dimensional scale and therefore a composite will be based on a 4-item composite. These four items best reflect participants' confidence to self-regulate in the face of actual barriers, including exercising regularly in the face of bad weather, while on vacation, without encouragement, and when under personal stress. These four items will be averaged to generate our main outcome of interest, and the remaining nine items will be assessed for exploratory purposes.
Martial arts experience | Participants will be assessed once, at baseline.
  A novel questionnaire will assess prior martial arts experience. For example, "Do you have any experience with martial arts or combat training? This includes any combat training as part of military or police service." Individual item averages and frequencies will be used to describe the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Exercise, Technology, and Cognition Laboratory - Louise Freer Hall 284, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to the Primary investigator and Lead research assistant of this study.